CLINICAL TRIAL: NCT02368834
Title: Evaluation of a Psychoeducation Program for the Parents of Attention Deficit Hyperactivity Disorder
Brief Title: Psychoeducation for the Parents of Attention Deficit Hyperactivity Disorder (ADHD) Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Li Yang, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2011-4024-04-01
Record Dates: First submitted 2015-02-12; First posted 2015-02-23 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): A psychoeducation program was delivered to the parents/caregivers
  Interventions: Behavioral: psychoeducation
- control group (No Intervention): This group waited for 3 months, only receiving general consultation.

INTERVENTIONS:
Behavioral: psychoeducation — The intervention included a presentation by a psychiatrist, with parent manual provided, and then two group sessions at the 2nd and 4th weeks to address further concerns of the parents
  Arms: intervention group

SUMMARY:
This study designed and evaluated a psychoeducation program for parents of ADHD children in terms of improving medication adherence and clinical benefits.

DETAILED DESCRIPTION:
ADHD is the most common behavioral disorder with poor outcomes. Medication is the most important treatment for ADHD. The adherence to the medication is extremely low. This study aims to investigate the the effect of a psychoeducation program for parents of ADHD children. The investigators intent to recruit 80 ADHD families. They will be randomized to intervention group and control group using a block randomization design. The intervention group will participate in a psychoeducation program, which includes a presentation from a specialist in ADHD at the baseline, with parent manual provided, posters, and two group sessions at the end of the 2nd and the 4th weeks. The control group only receives general consultation. The knowledge towards ADHD and its treatment, parents' behavior intent, medication adherence, clinical symptoms, and parents' satisfaction will be assessed and compared at the end of the 1st and 3rd months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* parents of ADHD children diagnosed with ADHD
* 6 - 16 years old;
* first referral to the hospital;
* candidate for medication according to both the doctor and the family

Exclusion Criteria:

* inappropriate for medication;
* being illiterate of the parent or the primary caregiver;
* unable to be followed-up.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Medication adherence rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD, Principal Investigator — Peking University Sixth Hospital
Locations (1):
- Peking University Sixth Hospital, Beijing, Beijing Municipality, China